CLINICAL TRIAL: NCT02945852
Title: Phase II Study of Apatinib as Third- or Further-line Treatment for Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Apatinib for Extensive Stage Small Cell Lung Cancer After Second/Third Line Chemotherapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fan Yun, MD (Other)
Responsible Party: Sponsor-Investigator, Fan Yun, MD, Doctor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zjSAPA001
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib

ARMS (1):
- refractory SCLC (Experimental): Patients receive apatinib 500mg/d until progressive Disease(PD).
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: apatinib — apatinib 500mg/d until progressive Disease

SUMMARY:
Although fist-line therapy with Cisplatin and etoposide(EP)or Carboplatin and etoposide(CE)and second-line therapy with topotecan has been given, patients with extensive small cell lung cancer(ED-SCLC) still relapse and 2-year survival is less than 10%. There is no standard treatment recommendation for this group of patients who failed to second-line therapy and had good performance status. Apatinib has been approved as a second-line treatment for advanced gastric cancer. Several phase III clinical studies of non small cell lung cancer, liver cancer, colorectal cancer and other tumors also showed apatinib has less toxic side effects and better patient tolerance. However, the clinical application of apatinib in small cell lung cancer is still lack of evidence-based medicine. And this clinical trial is designed to prospectively investigate the efficacy and safety of apatinib in refractory or recurrent ED-SCLC patients in our center.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is a highly aggressive disease characterized by its rapid doubling time, high growth fraction, early development of disseminated disease, and dramatic response to first-line chemotherapy and radiation. Small cell lung cancer accounts for approximately 20%-25% lung cancer patients. SCLC patients are categorized as limited disease, defined as disease that is confined to the ipsilateral hemithorax that can be encompassed within a tolerable radiation port, or extensive disease (ED), defined as the presence of overt metastatic disease determined by imaging or physical examination. Two third of patients are diagnosed with ED at presentation. Despite the development of novel cytotoxic drugs, the therapeutic approach to SCLC has been stagnant for more than twenty years. Standard treatment for ED-SCLC remains EP or CE, a regimen that yield a median survival of approximately 9 months and a 5-year survival of less than 1%.In some guidelines for SCLC, topotecan is recommended as the standard second-line treatment in patients who relapse less than 3 months. As for patients who relapse more than six months after the end of initial treatment, EP or CE regimen is recommended to be used again.There is no standard treatment recommendation for this group of patients who failed to second-line therapy.Apatinib has been approved as a second-line treatment for advanced gastric cancer. Several phase III clinical studies of non small cell lung cancer, liver cancer, colorectal cancer and other tumors also showed apatinib has less toxic side effects and better patient tolerance.And this clinical trial is designed to prospectively investigate the efficacy and safety of apatinib in refractory or recurrent ED-SCLC patients.

ELIGIBILITY:
Inclusion Criteria:

Histologic or cytologic diagnosis of small cell lung caner(SCLC), Extensive Stage.

Previous treatments including first-line therapy with EP or CE and second-line therapy with topotecan; Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2; Males or females between 18 Years to 75 Years. Expected survival is above three months. At least one measurable lung tumor lesion (according to RECIST criteria, the application of conventional technology, diameter length of the lesion >= 20mm or spiral CT >=10mm).

Adequate hematologic (Leukocyte count >= 4.0×109/L, neutrophil count>=2.0×109/L, hemoglobin>=95g/L, platelets>=100×109/L), hepatic function (aspartate transaminase (AST) & alanine transaminase(ALT) =<upper normal limit(UNL) x1.5, bilirubin level =< UNL x 1.5).

Patient can take oral medicine. Patients have the ability to understand and voluntarily sign the informed consent, and allow adequate follow-up.

Exclusion Criteria:

History of cardiovascular disease: congestive heart failure (CHF) > New York Heart Association (NYHA) II, active coronary artery disease(patients with myocardial infarction six months ago can be recruited), arrhythmias need to be treated (allow taking beta blockers or digoxin).

Serious clinical infection (> NCI-CTCAE version 4.0 ,infection standard II). Patients with epilepsy who need to take medicine (such as steroids or anti epilepsy agents).

The patients had accepted allogeneic organ transplantation. Bleeding tendency or coagulation disorders. Patients who need renal dialysis. Suffered from other tumor within 5 years( Except: cervical carcinoma in situ, cured basal cell carcinoma, cured bladder epithelial tumor).

Uncontrolled hypertension (systolic pressure>150 mmHg , or diastolic pressure> 90 mmHg).

Thrombosis or embolism(cerebrovascular accidents including transient ischemic attack within the last 6 months).

Pulmonary hemorrhage >CTCAE grade 2 within 4 weeks before first use of drugs. Other organ hemorrhage >CTCAE grade 3 within 4 weeks before first use of drugs. severe uncured wounds, ulcers or fracture. uncured dehydration. Factors influencing the safety and compliance of patients. Inability to comply with protocol or study procedures. Pregnant or breast-feeding. The researcher believe that the Patient is not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-05-26 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 3 months
  The first day of treatment to the date that disease progression is reported.

SECONDARY OUTCOMES:
Tumor response rate | 3 months
  The ratio between the number of responders and number of patients assessable for tumor response.
Treatment-related adverse events | 3 months
  Treatment-related adverse events are assessed by common terminology criteria for adverse events(CTCAE) V4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Xu Y, Huang Z, Lu H, Yu X, Li Y, Li W, Chen J, Chen M, Gong L, Chen K, Qin J, Xu X, Jin Y, Zhao J, Shi X, Han N, Xie F, Zhang P, Xu W, Fan Y. Apatinib in patients with extensive-stage small-cell lung cancer after second-line or third-line chemotherapy: a phase II, single-arm, multicentre, prospective study. Br J Cancer. 2019 Oct;121(8):640-646. doi: 10.1038/s41416-019-0583-6. Epub 2019 Sep 16. PMID 31523058